CLINICAL TRIAL: NCT01943604
Title: The Effects of Breakfast on Neuropsychological Functioning in Children Ages 8-10 From Low to Middle Income Families
Brief Title: The Effects of Breakfast on Neuropsychological Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Ferrero Italy, Inc. (Industry)
Responsible Party: Principal Investigator, Theresa A Nicklas, Professor, Baylor College of Medicine
Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-28698
Record Dates: First submitted 2013-08-08; First posted 2013-09-17 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Neuropsychology
Keywords: Neuropsychology; Breakfast eating patters; Glucose; Child Psychology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Nutella Breakfast
  Waffle Breakfast
  Interventions: Other: Nutella Breakfast; Other: Waffle Breakfast

INTERVENTIONS:
Other: Nutella Breakfast — Breakfast composed of bread and Nutella, milk and apple slices
Other: Waffle Breakfast — Breakfast composed of waffles and syrup, milk, and apple slices

SUMMARY:
This study is designed to examine healthy children who skip breakfast and the effects of fasting on their neuropsychological functioning and the potential benefits that a Balanced Breakfast may have on their learning abilities. It is expected that this study will provide new knowledge on how prolonged periods of 8 or more hours without food affect neurocognitive processes and thus learning how specific meals following this period of fasting, which most children experience, change those processes, potentially for the better.

The hypotheses for this study are:

1. Children who consume breakfast will demonstrate significantly higher levels of attention, greater concentration, and diminished impulsivity compared to children who do not consume breakfast.
2. Children who consume breakfast will demonstrate a significantly quicker reaction time and increased accuracy in correctly identifying target stimuli from an array compared to children who do not consume breakfast.
3. Children who consume breakfast will demonstrate increased freedom from distractibility and enhanced short-term memory compared to children who do not consume breakfast.
4. Children who consume breakfast will demonstrate increased cognitive processing speed compared to children who do not consume breakfast.
5. Children who consume breakfast will have improved verbal learning compared to children who do not consume breakfast.
6. Children who consume breakfast will have improved visual memory compared to children who do not consume breakfast.

DETAILED DESCRIPTION:
Hunger can be considered a chronic health condition. Among children, the lack of available food to meet usual physical needs on a regular basis leads to poor cognitive and behavioral performance and is associated with adverse physical and mental health outcomes. All of these findings are well documented among poor children living in families with sufficient food and are exacerbated even more among those in families living under conditions of food insufficiency. There has been a significant effort over the past 2 decades to document the effects of mechanisms of how hunger affects learning, cognitive performance, and behavior and how a meal, such as breakfast can mitigate those effects.

The longest period during a 24-hour day when children go without food is the period from the beginning of sleep at night to the first meal of the following day. Therefore, the morning seems an ideal time to examine those biological factors that result from hunger or fasting and how they affect basic processes that underpin learning and behavior. Underprivileged but otherwise healthy children seem most affected by hunger. Thus, studies are needed to compare children from families of different economic income strata to understand better how a breakfast meal might affect those learning and behavioral processes, and whether the breakfast meal truly has a positive effect on basic learning and behavior.

The goal of this study is to evaluate the effects on short-term neuropsychological functioning of: a) consumption of breakfast versus no breakfast (2 different breakfast meals will be employed); and b) consumption of breakfast by groups of children from low income families vs children from families with average/middle incomes, who are 8-10 years of age. The primary outcome will be neuropsychological functioning in specific areas of cognition, as measured by standardized tests. A secondary outcome will be glucose homeostasis, measured by blood ketones and blood glucose and insulin.

A total of 154 children will be recruited with an anticipated 20% drop out rate. The final sample will consist of 64 children in each socioeconomic group (total n=128) who will stay overnight three separate nights and participate in each breakfast condition. The sample will consist of low and middle income African- and Hispanic-Americans and Caucasian male and female children between the ages of 8-10. The sample size will consist of an equal number of boys and girls and will have an equal representation of children from the socioeconomic conditions (i.e. low and middle income) and ethnicities (African and Hispanic Americans and Caucasians) identified.

The design consists of two independent groups based on SES with a crossover, repeated-measures (within subject and across subject design, under three breakfast conditions. The outcome measures (dependent variables) will include a battery of neuropsychological measures. All participating subjects are admitted to the Children's Nutrition Research Center (CNRC) Metabolic Research unit (MRU) three times for overnight stays with intervals of at least 2 weeks apart across 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-10 years of age will be recruited from Houston, Texas
* Low socio-economic (SES) children and middle income children (defined as those who receive "free" and "reduced fee" lunches from the respective schools within the district)

Exclusion Criteria:

* Children with weights below the 10th percentile and above the 90th percentile will be excluded
* Children will be examined by a trained nurse to rule out color blindness
* Children with a history of neurological, neurodevelopmental, developmental learning disabilities, sensory impairments, mood disorders, attention deficit hyperactivity disorder, acute or chronic medical conditions, reported lactose intolerance, veganism, asthma, tree nut and/or peanut allergy, anemia, pubescent, on prescription medications or a Tanner stage greater than 2 will be excluded from the study
* Subjects who are unwilling to consume Nutella or have dietary restrictions that would prevent them from consuming the prepared meals will not be included

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visual Search Paradigm change across three timepoints | Administered three times across three months
  The Padova Visual Search Paradigm will be used to assess sustained attention. This measure requires the participant to make a decision about the presence of a specified target object in an array of simultaneously presented objects. Stimulus generation and response recording will be conducted by a software package E-Prime 2.0 and running on a Pentium PC connected to a 13-inch screen. The protocol developed by Padova for children will be used in this study.
CPT-II change across three timepoints | Administered three times across three months
  A normed computerized test designed to assess attention, vigilance, and impulsivity. Reaction times and accuracy are also calculated. This measure takes 14 minutes to complete and can be administered to individuals ranging in age from 6 years old to 55+ years. This task involves the subjects sitting in front of a computer screen while letters of the alphabet are flashed briefly, at various inter-stimulus intervals. The subject is instructed to press the spacebar on the keyboard whenever a letter is seen on the screen, except the letter "X". The CPT-II will also be used to examine the correlation with the experimental visual search measure, and possibly offer external validity.
WISC-IV subtests (Working Memory/Attention) change across three timepoints | Administered three times across three months
  The Wechsler Intelligence Scale for Children-IV (WISC-IV) is an individually administered, comprehensive clinical instrument designed to assess intellectual functioning in children ages 6 years, 0 months to 16 years, 11 months.
  1. Digit Span - this subtest is composed of 2 parts, Digit Span Forward and Digit Span Backwards. This subtest is designed as a measure of auditory short-term memory, sequencing skills, attention, and concentration (Sattler, 2001). Each of the 2 parts of this subtest involves different discrete areas of cognition.
  2. Letter-Number Sequencing - this subtest is one of the core Working Memory Composite tests. The subject is provided a sequence of numbers and letters, and is asked to recall the numbers in descending order and the letters in alphabetical order.
WRAML2 subtests change across three timepoints | Administered three times across three months
  The Wide Range Assessment of Memory and Learning- Second Edition (WRAML 2) is a battery of subtests designed to examine the memory abilities in individuals ages 5 to over 85. The subtests to be administered in this study are the following :
  1. The Verbal Learning subtest - The task evaluates a person's ability to actively learn unrelated verbal material. For subjects ages 8 years and younger, 13 words are used. For subjects 9 years and older, 16 words make up this list-learning tasks. A subtest Scale Score is obtained based on the total number of words remembered correctly on the 4 learning trials.
  2. The Picture Memory subtest - is a test designed to assess visual memory.
TOMAL subtest change across three timepoints | Administered three times across three months
  The Test of Memory and Learning (TOMAL) is a comprehensive memory battery standardized for use with children and young adults.
  a) Visual Selective Reminding (VSR) - is a nonverbal analog to the Word Selective Reminding (WSR) subtest of the TOMAL. The subjects are required to point to specified dots on a card, following a demonstration by the examiner, and are reminded only of the items recalled incorrectly. Trials continue until mastery is achieved or until 8 trials have been attempted. It is designed to assess learning and immediate recall functions of visual (nonverbal) memory.
WISC-IV subtests (Processing Speed) change across three timepoints | Administered three times across three months
  For each of the subtests, the distribution of each age group's total raw scores is converted to scaled scores with a mean of 10 and a standard deviation (SD) of 3.
  1. Coding - In addition to cognitive processing speed, the subtest measures/involves short-term memory, learning ability, visual perception, visual-motor coordination, visual scanning ability, cognitive flexibility, attention, and motivation (Sattler, 2001).
  2. Symbol Search - In addition to processing speed, the subtest also involves short-term visual memory, visual-motor coordination, cognitive flexibility, visual discrimination, and concentration (Sattler, 2001).

SECONDARY OUTCOMES:
Blood Ketones | Blood draws occur before and after each breakfast treatment and neuropsychological testing for a total of 6 blood draws across 3 months
  Blood Ketones (e.g. beta-hydroxybutyrate) will be measured on collected blood samples. Ketone measurements will allow us to determine if the children have depleted their glucose stores during the overnight fast to the point that they are metabolizing fat for energy.
Demographic Questionnaire | Administered one time across three months
  A demographic questionnaire will be used to document age, ethnicity, gender, and socioeconomic status and to verify whether the child receives free/reduced price/paid lunches. The socioeconomic portion of the questionnaire comes from the same questionnaire used by the National Poverty Center for calculation of poverty thresholds and whether the family income is at or below the national poverty level.
Breakfast Consumption Patterns | Administered one time across three months
  A short survey will be conducted to determine the frequency and quality of breakfast typically consumed.
Food Insecurity Scale | Administered one time across three months
  The Children's Food Security Scale will be used to measure the level of food security for the study subject and is calculated from the response to eight questions that ask specifically about food-related experiences and conditions of children. The scale measures the severity of food insecurity among children in surveyed households and identifies- in the most severe range of the scale- households in which children have been hungry at times because of a lack of household resources for food.
Children's Sleep Habits Questionnaire (CSHQ) | Administered one time across three months
  This measure will be used to determine if subjects have experienced sleep disturbances that may affect their performance on the neuropsychological tests. The CSHQ is a retrospective, 33-item parent questionnaire is the same is used in a number of studies to examine sleep behavior in young children. The CSHQ includes items relating to a number of key sleep domains that encompass the major presenting clinical sleep complaints in this age group: bedtime behavior and sleep onset; sleep duration; anxiety around sleep; behavior occurring during sleep and night waking; sleep-disordered breathing; parasomnias; and morning waking/daytime sleepiness. Parents are asked to recall sleep behaviors occurring over a "typical" recent week. Items are rated on a three-point scale: "usually" if the sleep behavior occurred five to seven times/week; "sometimes" for two to four times/week; and "rarely" for zero to one time/week.
Family Inventory of Life Events and Changes (FILE) Questionnaire | Administered one time across three months
  The FILE will be used to determine if subjects have experienced unusually high levels of family stress that may affect their performance on the neuropsychological tests. The FILE assesses the combined effects of life events experienced by a family and was developed as an index of family stress. The FILE is a 71 item self-report measure which is designed to record the normative and non-normative life events and changes experienced by a family unit in the past year. There are nine factor structures for FILE: 1) intra-family strains conflict, 2) marital strains, 3) pregnancy or childbearing strains, 4) finance and business strain, 5) work-family transitions and strains, 6) illness and family "care" strains, 7) losses, 8) transitions "in and out", and 9) family legal violations. Procedures have been established to generate a total stress score.
Physical Exam | Administered one time across three months
  Routine history and physical exam will be conducted by a physician. Height, weight, and assessment of Tanner stage, vital signs, and other routine examinations will be conducted. This exam also serves as a screening measure (e.g., history of drugs, developmental issues) that may affect participation status.
Blood measurements | Blood draws occur before and after each breakfast treatment and neuropsychological testing for a total of 6 blood draws across 3 months
  Serum glucose and insulin levels will be determined two times during each stay: on awakening and after neuropsychological testing. We are looking to see if there is a correlation between serum glucose levels and neuropsychological functioning at an age when the brain is taking up more glucose per kg of brain and body weight than later in life and therefore the child is potentially more vulnerable to the effects of low blood glucose. The insulin levels are done to determine if insulin responses are appropriate for the measured glucose levels or if they are responsible for the observed glucose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Nicklas, DrPH, Principal Investigator — Baylor College of Medicine; Isabella Iovino, PhD, Principal Investigator — Baylor College of Medicine; Janice Stuff, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Iovino I, Stuff J, Liu Y, Brewton C, Dovi A, Kleinman R, Nicklas T. Breakfast consumption has no effect on neuropsychological functioning in children: a repeated-measures clinical trial. Am J Clin Nutr. 2016 Sep;104(3):715-21. doi: 10.3945/ajcn.116.132043. Epub 2016 Jul 27. PMID 27465375